CLINICAL TRIAL: NCT05405504
Title: Evaluation of ReDS Pro System V2.7 and ReDS ICU in Patients With Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Christian Hassager (Other)
Responsible Party: Sponsor-Investigator, Christian Hassager, MD, DMSc, Professor in Cardiology, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: HJE-REDS-0001
Record Dates: First submitted 2022-05-23; First posted 2022-06-06 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- ICU part: Acute heart failure patients with Swan-Ganz catheter and an arterial catheter.
  Interventions: Device: Remote Dielectric Sensing (ReDS)
- Out-patient part: Chronic heart failure patients with CardioMEMS.
  Interventions: Device: Remote Dielectric Sensing (ReDS)

INTERVENTIONS:
Device: Remote Dielectric Sensing (ReDS) — Non-invasive device designed for the measurement of lung fluid using extremely low power electromagnetic waves. The ReDS Pro System V2.7 system has CE approval (3900874CE01) and FDA clearance.

SUMMARY:
The study is an investigator-initiated, prospective cohort trial. The trial aims to evaluate ReDS Pro System V2.7 and ReDS ICU in patients with heart failure (HF).

DETAILED DESCRIPTION:
The study is an investigator-initiated, prospective cohort trial. The trial aims to evaluate ReDS Pro System V2.7 and ReDS ICU in patients with heart failure (HF). The overall purposes are:

* to evaluate the ReDS efficacy measurements of lung fluid compared to pulmonary artery pressure guided therapy with CardioMEMS in out-patients with HF.
* to describe the feasibility of ReDS ICU in patients admitted to an ICU with HF

For the out-patient part, the patients will be recruited from the outpatient clinic at Rigshospitalet. The patient must be at least 18 years, have a history of chronic HF, and already monitored using CardioMEMS and must not fulfill any of the exclusion criteria.

For the ICU part, the patients will be recruited at the ICU department at the Heart Center at Rigshospitalet. The patient must be at least 18 years, intubated, and unconscious or sedated (Glasgow Coma Score <8), and already monitored using Swan-Ganz and arterial catherization and must not fulfill any of the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

ICU part:

* at least 18 years of age
* hospitalized in ICU setting at Rigshospitalet
* intubated
* unconscious or sedated (Glasgow Coma Score <8)
* monitored using Swan-Ganz and arterial catherization.

Out-patient part:

* at least 18 years of age
* history of Chronic heart failure > 3 months
* CardioMEMS

Exclusion Criteria:

ICU part:

* pacemaker or ICD on the right side
* congenital heart malformations or intra-thoracic mass that would affect the right lung anatomy (e.g. dextrocardia, lung carcinoma)
* wounds, burns, healing tissue, skin infection or recent skin graft or flap where the sensors should be attached to the skin
* habitus is out of range due to one or more of the following
* height less than 155 cm or higher than 195 cm
* estimated BMI of less than 22 or more than 36
* standard active therapy has been stopped as the patient is inevitably dying.

Out-patient part:

* pacemaker or ICD on the right side
* congenital heart malformations or intra-thoracic mass that would affect the right lung anatomy (e.g. dextrocardia, lung carcinoma)
* wounds, burns, healing tissue, skin infection or recent skin graft or flap where the sensors should be attached to the skin
* habitus is out of range due to one or more of the following Height less than 155 cm or higher than 195 cm BMI of less than 22 or more than 38 For BMI 36 to 38, chest size ruler should be 39 or less
* cancer or other severe non-cardiac disease with estimated life expectancy less than 1 year
* planned hospitalization for ICD, pacemaker, lung or heart surgery including heart transplantation during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU part:
  Acute heart failure patients with Swan-Ganz catheter and an arterial catheter.
  Outpatient part:
  Chronic heart failure patients with CardioMEMS.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between ReDS ICU fluid parameters and Swan-Ganz measurements | Daily Swan-Ganz catheter and ReDS ICU measurements the first 72 hours after Swan-Ganz implantation
  Measurements on Swan-Ganz catheter (CVP, PAP, PCWP - all in mmHg) and the percentage of fluid in the lungs (%)
Correlation between ReDS v2.7 fluid parameters and CardioMEMS measurements | 3 months
  mPAP (mmHg), dPAP (mmHg) and the percentage of fluid in the lungs (%)

SECONDARY OUTCOMES:
Changes in ReDS ICU fluid parameters following changes in Positive End Expiratory Pressure | During the first 72 hours after Swan-Ganz implantation
  The percentage of fluid in the lungs (%) and PEEP
Changes in ReDS ICU fluid parameters following raised leg test | During the first 72 hours after Swan-Ganz implantation
  The percentage of fluid in the lungs (%)
Changes in ReDS ICU fluid parameters following changes in body position | During the first 72 hours after Swan-Ganz implantation
  The percentage of fluid in the lungs (%)
Changes in ReDS ICU fluid parameters following changes administration of diuretics and inotropic/inodilators | During the first 72 hours after Swan-Ganz implantation
  The percentage of fluid in the lungs (%)
Correlation between ReDS v2.7 fluid parameters and body weight | 3 months
  The percentage of fluid in the lungs (%)
Correlation between ReDS v2.7 fluid parameters and dyspnea symptom evaluated by NYHA class. | 3 months
  The percentage of fluid in the lungs (%)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hassager, MD, DMSc, Professor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data is planned to be available upon reasonable request via the Principal Investigator pending final, complete publication of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Access and final IPD criteria is pending final, complete publication of the study.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA)

REFERENCES:
- [Background] Sattar Y, Suleiman A, Mir T, et al. TREND OF HEART FAILURE READMISSION PREVENTION IN REMOTE DIELECTRIC SENSING (REDS) MONITORING- A META-ANALYSIS. J Am Coll Cardiol. 2021 May, 77 (18_Supplement_1) 808.
- [Background] Abraham WT, Bensimhon D, Pinney SP, Feitell SC, Peacock WF, Amir O, Burkhoff D. Patient monitoring across the spectrum of heart failure disease management 10 years after the CHAMPION trial. ESC Heart Fail. 2021 Oct;8(5):3472-3482. doi: 10.1002/ehf2.13550. Epub 2021 Aug 13. PMID 34390219
- [Background] Amir O, Azzam ZS, Gaspar T, Faranesh-Abboud S, Andria N, Burkhoff D, Abbo A, Abraham WT. Validation of remote dielectric sensing (ReDS) technology for quantification of lung fluid status: Comparison to high resolution chest computed tomography in patients with and without acute heart failure. Int J Cardiol. 2016 Oct 15;221:841-6. doi: 10.1016/j.ijcard.2016.06.323. Epub 2016 Jul 1. PMID 27434357
- [Background] Uriel N, Sayer G, Imamura T, Rodgers D, Kim G, Raikhelkar J, Sarswat N, Kalantari S, Chung B, Nguyen A, Burkhoff D, Abbo A. Relationship Between Noninvasive Assessment of Lung Fluid Volume and Invasively Measured Cardiac Hemodynamics. J Am Heart Assoc. 2018 Nov 20;7(22):e009175. doi: 10.1161/JAHA.118.009175. PMID 30571493
- [Background] Lala A, Barghash MH, Giustino G, Alvarez-Garcia J, Konje S, Parikh A, Ullman J, Keith B, Donehey J, Mitter SS, Trivieri MG, Contreras JP, Burkhoff D, Moss N, Mancini DM, Pinney SP. Early use of remote dielectric sensing after hospitalization to reduce heart failure readmissions. ESC Heart Fail. 2021 Apr;8(2):1047-1054. doi: 10.1002/ehf2.13026. Epub 2020 Dec 18. PMID 33336881
- [Background] Amir O, Rappaport D, Zafrir B, Abraham WT. A novel approach to monitoring pulmonary congestion in heart failure: initial animal and clinical experiences using remote dielectric sensing technology. Congest Heart Fail. 2013 May-Jun;19(3):149-55. doi: 10.1111/chf.12021. Epub 2013 Jan 25. PMID 23350643
- [Background] Bensimhon D, Alali SA, Curran L, Gelbart E, Garman DWV, Taylor R, Chase P, Peacock WF. The use of the reds noninvasive lung fluid monitoring system to assess readiness for discharge in patients hospitalized with acute heart failure: A pilot study. Heart Lung. 2021 Jan-Feb;50(1):59-64. doi: 10.1016/j.hrtlng.2020.07.003. Epub 2020 Jul 20. PMID 32703623
- [Background] Imamura T, Hori M, Koi T, Fukui T, Oshima A, Fujioka H, Ueno Y, Onoda H, Tanaka S, Fukuda N, Ueno H, Kinugawa K. Relationship Between Body Posture and Lung Fluid Volume Assessed Using a Novel Noninvasive Remote Dielectric Sensing System. Circ Rep. 2021 Dec 3;4(1):25-28. doi: 10.1253/circrep.CR-21-0130. eCollection 2022 Jan 7. PMID 35083385
- [Background] Amir O, Ben-Gal T, Weinstein JM, Schliamser J, Burkhoff D, Abbo A, Abraham WT. Evaluation of remote dielectric sensing (ReDS) technology-guided therapy for decreasing heart failure re-hospitalizations. Int J Cardiol. 2017 Aug 1;240:279-284. doi: 10.1016/j.ijcard.2017.02.120. Epub 2017 Mar 3. PMID 28341372

DOCUMENTS (1):
  • Study Protocol (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT05405504/Prot_000.pdf